CLINICAL TRIAL: NCT06766279
Title: Investigating the Efficacy of OMT to Recover Olfactory Perception After COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burrell College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Thomas Eiting, Assistant Professor of Physiology, Burrell College of Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0118_2023
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Anosmia
MeSH Terms: conditions — Anosmia | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OMT (Experimental): Subjects will undergo an evaluation of their sense of smell using a thoroughly-vetted and published protocol. If subjects are found to have a reduced sense of smell, they will be assigned to either the OMT or sham intervention. The OMT intervention will consist of two procedures: occipitoatlantal decompression and treating the nasal Chapman point. Subjects will then be evaluated after receiving treatment, as well as a follow-up visit the day after, and a final visit within 1-2 weeks post treatment.
  Interventions: Procedure: Osteopathic Manipulative Treatment
- Sham (Sham Comparator): Subjects will undergo an evaluation of their sense of smell using a thoroughly-vetted and published protocol. If subjects are found to have a reduced sense of smell, they will be assigned to either the OMT or sham intervention. The sham intervention will consist of the experimenter resting their hands on the sides of the subject's neck. Subjects will then be evaluated after receiving treatment, as well as a follow-up visit the day after, and a final visit within 1-2 weeks post treatment.
  Interventions: Procedure: Sham treatment

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — The OMT intervention in this study will be comprised of an occipitoatlantal (OA) decompression and treatment of the nasal Chapman point. The OA decompression will be applied for 2 minutes with 12N of pressure as this pressure has been determined to produce the greatest effect. Treatment at this level reduces congestion of nasal mucosa. The suboccipital decompression technique is generally considered to bear minimal risks and is perceived by most patients as a pleasant experience. This technique is considered to be a basic skill among osteopathic physicians. It is usually taught within the first semester of the first year at Colleges of Osteopathic Medicine.
  The other intervention technique will be addressing the nasal Chapman points that are found at the tip of the transverse process of C1 and the costochondral junction of the first rib on each side. Both techniques are performed while the subject is supine.
  Arms: OMT
Procedure: Sham treatment — The sham intervention will consist of the subject lying supine with the investigator's hands resting gently on both sides of subject's neck for 5 minutes.
  Arms: Sham

SUMMARY:
One of the most widespread symptoms of COVID-19 is loss of the sense of smell. There are very few treatments for helping individuals recover their sense of smell. Osteopathic manipulative treatment (OMT) may be a useful tool in helping people recover their smell perception. In this study the investigators test whether OMT can be used to help individuals recover their sense of smell if they lost it during COVID-19.

DETAILED DESCRIPTION:
Objectives: The objective of this study is to determine if osteopathic manipulative treatment affects the sense of smell after COVID-19 infection. A secondary objective of this study is to determine how long the improvement in the sense of smell lasts.

Background and Hypothesis: One of the most widespread symptoms of COVID-19 is the substantial reduction (hyposmia) or complete loss of the sense of smell (anosmia) in affected individuals. Individuals who experience loss of smell report reductions in many metrics of quality of life (e.g., enjoyment of coffee or food), as well as facing a slight elevated risk of serious, life-threatening scenarios (e.g., delayed detection of smoke from fire). Some people who experience loss of smell experience a complete recovery concomitant with overall COVID-19 recovery. More commonly, however, is some degree of persistent loss of smell. In extreme cases individuals lose their sense of smell completely or retain only the most rudimentary of sensory abilities. Additionally, partial or complete loss of smell has emerged as an early and common symptom of Alzheimer's disease and other dementias, including dementias associated with Parkinson's disease. Whether the loss of smell from infections or allergies contributes to the risk of developing these conditions is unknown. The treatment for anosmia ranges from intranasal budesonide to stellate ganglion blockade. Little has been published regarding the use of osteopathic manipulative treatment (OMT) to treat anosmia in post-COVID-19 patients. The techniques that have been employed are advanced skills that few osteopathic physicians possess.

In this project, the investigators explore the possibility of employing (OMT) to help individuals recover some or all of their olfactory ability after a COVID-19 infection. The investigators will employ techniques that are commonly used in OMT to alleviate symptoms associated with sinusitis or other complaints associated with the nasal sinuses and airway. Specifically, the investigators have chosen to investigate the use of occipitoatlantal decompression and treatment of the Chapman nose point in providing relief from COVID-19 symptoms, because of their effectiveness in OMT for other nasal-related diseases or infections, their relative ease of use and of teaching to osteopathic medical students, who will be recruited as student investigators to contribute to this study and future studies for which the current proposal is laying the groundwork.

Study Subjects: All subjects will be adult (minimum age of 18 years) individuals of both genders who have tested positive for COVID-19. After an initial screening of their sense of smell, subjects who are found to have a normal odor identification ability will be excluded from the study.

Recruitment of Subjects: Subjects will be recruited from the Las Cruces community by word of mouth, as well as through the use of a simple flyer that will be generated and passed out to community members and posted on public message boards. The investigators will work with the Burrell College Office of Marketing and Public Relations to further devise a strategy for recruiting participants.

Number of Subjects: 32

Power Analysis: Please see Item 7.

Inclusion criteria: Minimum of 18 years of age, verified by an official picture ID, positive COVID-19 test with recent COVID-19 symptoms.

Exclusion criteria: Age under 18 years; pregnancy; any findings on the osteopathic screening/evaluation that would hinder the effectiveness or increase the risk associated with OA decompression; any medication that interferes with the sense of smell (intranasal zinc, intranasal antihistamines, intranasal corticosteroids), allergic rhinitis, use of oral corticosteroids, antihistamines.

Consent and Enrollment: Prior to enrollment in the study, potential subjects will review the purpose of the study, eligibility for inclusion in the study (based on exclusion criteria listed above), potential risks and benefits, and the consent form with one of the researchers. Once written consent is obtained, the subjects will be asked to fill out a questionnaire that is designed to verify that the subject qualifies for inclusion in the study (based on exclusion criteria) and to obtain contact data (name, address, phone, e-mail) and demographic information (age, sex). Potential subjects may be excluded based on answers in the questionnaire. Each subject will be assigned a subject number that will be used to de-identify data.

Consent will also be obtained from the PI, co-PI, and student investigators as there is a possible risk of contracting COVID-19 despite wearing masks. Vaccination against COVID-19 will be recommended.

Study Subjects:

Decision on enrollment: The final decision on enrollment based on these criteria will be done by the PI, Dr. Eiting or the co-investigator, Dr. Kania.

Experimental Protocol: The general procedure for this study is as follows. The investigators will recruit subjects with and without a current COVID-19 infection, and ask them to undergo an olfactory behavioral test to determine their current olfactory acuity. Subjects with current COVID-19 infection will have evidence of a positive test, and will be evaluated not sooner than the sixth day of symptoms. The New Mexico Department of Health recommends quarantining for five days after the onset of symptoms of Covid infection. Investigators and subjects will wear masks covering their nose and mouth during evaluation and undergoing the interventions. After consent is obtained, subjects will be randomly assigned to the treatment or sham arms of the study. All subjects will undergo evaluation of their sense of smell via an olfactory test. The investigators will use the "Sniffin' Sticks" olfactory test, which has been validated and utilized in many scientific studies. The testing will be done in an open-air, well-ventilated room on the Burrell main campus. Subjects will then undergo OMT intervention or sham treatment (participants will not know to which group they are assigned), and their olfactory acuity will be tested again, post-intervention. An interval of at least one hour will be used between pre- and post-treatment olfactory testing. Subjects will be invited back to undergo olfactory testing again on a daily basis for up to 10 days. This is to determine the effectiveness of a single OMT intervention and how long the effect lasts, or the rate of spontaneously returned sense of smell.

The OMT intervention in this study will be comprised of an occipitoatlantal (OA) decompression and treatment of the nasal Chapman point. The OA decompression will be applied for 2 minutes with 12N of pressure as this pressure has been determined to produce the greatest effect. Treatment at this level reduces congestion of nasal mucosa. The suboccipital decompression technique is generally considered to bear minimal risks and is perceived by most patients as a pleasant experience. This technique is considered to be a basic skill among osteopathic physicians. It is usually taught within the first semester of the first year at Colleges of Osteopathic Medicine. There has been no untoward effects on students performing or receiving this technique in the fourteen years that the PI has taught the technique at BCOM or RVU-COM. She has not had any patients have adverse reactions to this technique during the nearly thirty years she was in practice.

The other intervention technique will be addressing the nasal Chapman points that are found at the tip of the transverse process of C1 and the costochondral junction of the first rib on each side. These techniques are safe and easily performed. Dr. Kania has extensive experience in teaching these techniques and training osteopathic medical students to perform them consistently for various studies.12 Both techniques are performed while the subject is supine.

Osteopathic manipulation is well-tolerated in general according to a study by Degenhardt et al., that found that only 45 out of 1847 visits for osteopathic manipulative treatment resulted in pain or discomfort, tiredness, fatigue, lightheadedness, nausea/vomiting, headache, numbness/tingling or stiffness following osteopathic treatment.

The sham intervention will consist of the subject lying supine with the investigator's hands resting gently on both sides of subject's neck for 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID-19 test or diagnoses
* Self-reported deficiency in sense of smell

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Any findings on the osteopathic screening/evaluation that would hinder the effectiveness or increase the risk associated with OA decompression
* Any medication that interferes with the sense of smell (intranasal zinc, intranasal antihistamines, intranasal corticosteroids)
* Allergic rhinitis
* Use of oral corticosteroids or antihistamines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Ability to Recover Sense of Smell after OMT | from enrollment until 2 weeks post treatment
  Data from 32 COVID-19-positive individuals will be collected. This group will be divided into 2 groups of 16: one of these groups will be given the OMT intervention, and one will be given a sham intervention. The sample size of 16 per group comes about as follows. The main dependent variable measured for each person will be the number of odors identified out of a panel of 16 odors. This will be in the form of a multiple-forced-choice questionnaire: participants will be required to identify the odor from a selection of possible options. Upon treatment and re-testing, we will measure the number of odors identified again. Previous work (Whitcroft et al. 2016, Rhinology 54:368-373) that has looked at the effects of sodium citrate treatment on odor identification ability has shown a mean improvement of just over 2 points using this same identification test (for example, subjects able to correctly identify 14 odors posttreatment and just 12 odors pre-treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Burrell College of Osteopathic Medicine, Las Cruces, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
An explicit plan to share these data has not been developed. We will share deidentified data as required by any journal in which we may publish the data collected for this project. We may revisit this plan in the future.

REFERENCES:
- [Background] Degenhardt BF, Johnson JC, Brooks WJ, Norman L. Characterizing Adverse Events Reported Immediately After Osteopathic Manipulative Treatment. J Am Osteopath Assoc. 2018 Mar 1;118(3):141-149. doi: 10.7556/jaoa.2018.033. PMID 29480914
- [Background] Kania AM, Weiler KN, Kurian AP, Opena ML, Orellana JN, Stauss HM. Activation of the cholinergic antiinflammatory reflex by occipitoatlantal decompression and transcutaneous auricular vagus nerve stimulation. J Osteopath Med. 2021 Feb 24;121(4):401-415. doi: 10.1515/jom-2020-0071. PMID 33694358
- [Background] Hummel T, Sekinger B, Wolf SR, Pauli E, Kobal G. 'Sniffin' sticks': olfactory performance assessed by the combined testing of odor identification, odor discrimination and olfactory threshold. Chem Senses. 1997 Feb;22(1):39-52. doi: 10.1093/chemse/22.1.39. PMID 9056084
- [Background] 8. Dostálová N. 2022. Effect of Osteopathic treatment on the post-covid loss of smell and taste. Thesis for Master of Science in Osteopathy, London College of Osteopathy and Health Sciences
- [Background] Jacob B, Sawhney M, Sridhar A, Jacob B, Muller J, Abu-Sbaih R, Yao SC. Potential therapeutic effects of adjunct osteopathic manipulative treatments in SARS-CoV-2 patients. J Osteopath Med. 2023 Apr 21;123(7):343-349. doi: 10.1515/jom-2022-0207. eCollection 2023 Jul 1. PMID 37079451
- [Background] Moon HS, Chon JY, Lee SH, Ju YM, Sung CH. Long-term Results of Stellate Ganglion Block in Patients with Olfactory Dysfunction. Korean J Pain. 2013 Jan;26(1):57-61. doi: 10.3344/kjp.2013.26.1.57. Epub 2013 Jan 4. PMID 23342209
- [Background] Nguyen TP, Patel ZM. Budesonide irrigation with olfactory training improves outcomes compared with olfactory training alone in patients with olfactory loss. Int Forum Allergy Rhinol. 2018 Sep;8(9):977-981. doi: 10.1002/alr.22140. Epub 2018 Jun 14. PMID 29901865
- [Background] Sun GH, Raji CA, Maceachern MP, Burke JF. Olfactory identification testing as a predictor of the development of Alzheimer's dementia: a systematic review. Laryngoscope. 2012 Jul;122(7):1455-62. doi: 10.1002/lary.23365. Epub 2012 May 2. PMID 22552846
- [Background] Domellof ME, Lundin KF, Edstrom M, Forsgren L. Olfactory dysfunction and dementia in newly diagnosed patients with Parkinson's disease. Parkinsonism Relat Disord. 2017 May;38:41-47. doi: 10.1016/j.parkreldis.2017.02.017. Epub 2017 Feb 21. PMID 28242255
- [Background] Cooper KW, Brann DH, Farruggia MC, Bhutani S, Pellegrino R, Tsukahara T, Weinreb C, Joseph PV, Larson ED, Parma V, Albers MW, Barlow LA, Datta SR, Di Pizio A. COVID-19 and the Chemical Senses: Supporting Players Take Center Stage. Neuron. 2020 Jul 22;107(2):219-233. doi: 10.1016/j.neuron.2020.06.032. Epub 2020 Jul 1. PMID 32640192
- [Background] Whitcroft KL, Hummel T. Olfactory Dysfunction in COVID-19: Diagnosis and Management. JAMA. 2020 Jun 23;323(24):2512-2514. doi: 10.1001/jama.2020.8391. No abstract available. PMID 32432682
- See also: COVID isolating — https://cv.nmhealth.org/archives/how-to-isolate-when-positive/